CLINICAL TRIAL: NCT04099693
Title: A Prospective Randomized Study of General Anesthesia Versus Anesthetist Administered Sedation for ERCP
Acronym: RAGE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King Abdullah Medical City (Other Government)
Responsible Party: Sponsor
Other Study IDs: 18-492
Record Dates: First submitted 2019-05-08; First posted 2019-09-23 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General Anesthesia: All the patients will be intubated and ventilated using cisatracurium (0.15 mg/kg) as a muscle relaxant and propofol (1.5-2mg/kg) for induction. The inhalational anesthetic, sevoflurane, will be used to maintain the depth of anesthesia using 50% mix of nitrous oxide and oxygen.
  Fentanyl will be used in both groups at a rate of 1-2 microgram /kg to achieve an adequate level of analgesia in both groups.
- Anesthetist Administered sedation for ERCP: To ensure a steady level of AAS each patient in this group will be sedated using propofol. An induction bolus of propofol (0.5 - 1 mg/kg) will be administered followed by continuous infusion with variable doses depending on the patients' age, weight, and clinical condition. In addition, fentanyl 1.5 μg/kg will be used at the anesthetist discretion.

SUMMARY:
Currently there no standard sedation techniques for performing ERCP. It is not clear whether sedation administered by anesthetist is better than anesthesia with intratracheal intubation. To clarify which of these sedative methods are better we plan to conduct a randomized trial comparing anesthetist administered sedation with general anesthesia in patients with ASA ≤3.

DETAILED DESCRIPTION:
ERCP is a relatively complex and lengthy endoscopic procedure. It is increasingly performed in elderly patients with multiple comorbidities and carries serious complications including death in about 0.33% of patients. An important aspect of endoscopy is sedation. The role of sedation is to make the procedure tolerable and acceptable to the patient by reducing anxiety and discomfort. It ensures that the patient is relatively still to avoid injury and enhance the chances of an efficient and successful procedure. Hence, adequate and appropriate sedation is of utmost importance to maximize patient comfort and minimize adverse events in ERCP.

The debate between anesthetist and gastroenterologist continues, as there is dearth of evidence evaluating the best form of sedative technique for ERCP.

Three prospective studies have tried to compare AAS with general anesthesia. Despite the fact that significantly more patients who had a higher body mass index (BMI) and were of ASA class 3 and above in the general anesthesia group, hypoxic events of less than 84% were much more common in patients having AAS then those who had general anesthesia (15% in AAS vs 6.7% in general anesthesia). On the other hand, hypotension (34% in general anesthesia vs 4% in AAS,) and arrhythmias (8% in general anesthesia vs 3% in AAS) were much more frequent in general anesthesia group than AAS. Upto 4% of patients had to be converted to general anesthesia due to cardiopulmonary compromise. However, the conclusion drawn was that AAS is as safe and effective as general anesthesia. Major caveats bring into question the conclusion. The studies were observational and non-randomized which introduces selection bias.

A recent randomized controlled trail that looked at general anesthesia versu AAS during ERCP concluded general anesthesia had a better safety profile than AAS (17). However, this study included only patient who were high risk for sedation related adverse events with ASA class >3 and the anesthesia was provided by nurse anesthetist. Hence, these results cannot be generalized. There are no randomized trials comparing AAS with general anesthesia in patients with ASA ≤3, which includes the vast majority of patients having ERCP

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Referred for ERCP
* Assessed by anesthetist
* ASA 1-3

Exclusion Criteria:

* Emergency situation (upper GI bleed, on mechanical ventilation)
* ASA class ≥4
* Distorted anatomy - like partial or total gastrectomy
* Pregnancy
* Unable to give or obtain consent and/ or disturbed level of consciousness
* Suspected difficult intubation using Ganzouri score > than 5 (18).
* Allergy to any study medication.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: all consecutive patients referred for ERCP who meet the below criteria will be approached to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 204 (Estimated)
Dates: Start 2019-09-08 (Actual); Primary Completion 2022-05-20 (Estimated); Study Completion 2022-05-20 (Estimated)

PRIMARY OUTCOMES:
The safety of anesthetist administered sedation (AAS) with general anesthesia for ERCP. | 2 years
  Significant cardiopulmonary complications will be defined as 1) Hypotension - when systolic BP drops below 25% of the baseline measurement requiring vasopressor drugs; 2) Cardiac Arrythmia - Bradycardia when heart rate drops below 50 beats/min or rises above 120 beats/min requiring treatment; 3) Hypoxia - when oxygen saturation falls below 90%; 4) Hypercapnia - when expiratory carbon dioxide increase by more than 25% from the baseline; 5) Apnea when respiratory activity ceases for ≥10 seconds via capnography; 6) Any interruption or termination of ERCP procedure related to sedation

SECONDARY OUTCOMES:
-The patient and endoscopist satisfaction with both types of sedation -The recovery time of AAS and general anesthesia | 2 years
  -Sedation induction time - the time from start of sedation till intubation of scope; - Procedure time - time from scope intubation till scope withdrawal; - Recovery time - time from scope withdrawal till recovery to healthy state scoring 10 on Aldrete system. - Success of ERCP - technical success of achieving deep cannulation of the ducts of interest in patients with native papillae without surgically altered anatomy; - Complications of ERCP - bleeding, perforation, pancreatitis.

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdullah Medical City, Holy Capital, Mecca, Makkah Western, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alzanbagi AB, Jilani TL, Qureshi LA, Ibrahim IM, Tashkandi AMS, Elshrief EEA, Khan MS, Abdelhalim MAH, Zahrani SA, Mohamed WMK, Nageeb AM, Abbushi B, Shariff MK. Randomized trial comparing general anesthesia with anesthesiologist-administered deep sedation for ERCP in average-risk patients. Gastrointest Endosc. 2022 Dec;96(6):983-990.e2. doi: 10.1016/j.gie.2022.06.003. Epub 2022 Jun 9. PMID 35690151